CLINICAL TRIAL: NCT03086967
Title: Cervical Ripening With a Double-lumen Balloon Catheter for Six Versus Twelve Hours
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-13-03B
Record Dates: First submitted 2017-02-21; First posted 2017-03-22 (Actual); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2017-03

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: cervical ripening; double lumen catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Six Hour (Active Comparator): Placement of foley catheter and extrusion after 6 hours followed by induction.
  Interventions: Device: Double-lumen balloon catheter
- Twelve Hour (Active Comparator): Placement of foley catheter and extrusion after 12 hours followed by induction.
  Interventions: Device: Double-lumen balloon catheter

INTERVENTIONS:
Device: Double-lumen balloon catheter — introduction of catheter into cervix for ripening prior to induction of labor following standard of care practices
  Other Names: foley bulb

SUMMARY:
The Foley catheter is a safe, effective method for cervical ripening. Limited data exists to indicate ideal time of placement for optimal cervical ripening prior to induction. The proposed study is a randomized control trial to determine if shortening placement from 12 to 6 hours of foley catheter can decrease time from start of induction to delivery. The prediction is that shortening foley bulb placement will result in shorter induction times, increased patient satisfaction and decreased length of stay on labor and delivery with secondary decreased medical costs.

DETAILED DESCRIPTION:
Objective: To determine whether a double-lumen balloon catheter requires twelve hours in the cervical canal to achieve its maximal cervical dilation. It is the hypothesis that the maximum cervical dilation and benefits of a double lumen foley catheter are achieved within the initial six hours after placement.

Study Design:

Overview: All eligible patients with a singleton pregnancy at 37 weeks gestational age or greater who are presenting for a clinically/ medically indicated induction with an unfavorable cervical exam will be invited to participate. As per the American College of Obstetricians and Gynecologists (ACOG) guidelines, all inductions performed prior to 39 weeks are medically indicated. Medical indications for induction prior to 39 weeks include but are not limited to preeclampsia, oligohydramnios and growth restriction. Upon admission to Labor and Delivery, women will be assessed for eligibility by an obstetric physician. A digital cervical examination will be performed and a Bishop score assigned. Patients with a Bishop score ≤ 6 are thought to benefit from a cervical ripening agent and the participants will be randomized based on parity at this point.

Type of Study: This study will be a prospective, randomized clinical control trial with human subjects.

Materials and Methods:

A qualified obstetric provider will provide eligible women with details of the study, including study objectives and methods. Consent will be obtained and witnessed from patients who elect to participate. Enrollment and randomization in the study will then occur. Patients will be randomized to the two groups using computer generated random numbers. The randomization will be stratified based on parity (i.e., women who have had any prior vaginal delivery above 20 weeks gestation v. women who have not). A foley bulb will then be placed by a qualified obstetric provider. Foley bulb will be inserted with or without speculum technique and with or without use of a stylet. In accordance with the standard of care, sterile saline will be placed in the intrauterine and vaginal balloon as tolerated by the patient for no more than a maximum of 80 cc in each balloon. The use of concomitant low dose pitocin with the foley bulb will be at the discretion of the admitting obstetric team. If the patient's foley bulb does not spontaneously expel within the maximum allotted time, they will be manually removed at six or twelve hours. At the time of manual removal or expulsion of the foley balloon, the patient's cervix will be checked by an experienced obstetric provider. As per usual protocol, additional cervical ripening and labor induction will proceed per managing obstetric team.

Independent Variables:

Data collection will include the independent variables of maternal age, parity, BMI, race (Caucasian, African American, Hispanic, Asian, other), Bishop Score, use of magnesium and epidural use. Data collection of independent fetal variables will include gestational age and estimated fetal weight.

Outcome Variables:

The primary outcome will be time from foley bulb placement to time of delivery. Secondary outcomes will include time from foley bulb placement to extrusion and rate of cesarean section. Additional comparison variables include: neonatal weight, APGAR scores and intrapartum and postpartum infection rates.

ELIGIBILITY:
Inclusion Criteria:

1. Intrauterine pregnancy at 37 weeks gestational age or greater as determined by best obstetrical dating criteria
2. Singleton gestation
3. Vertex presentation
4. Clinically adequate pelvis
5. Bishop Score less than or equal to 6
6. 16 years and older

   * North Carolina state law provides for the emancipation of minors, Chapter 7B-Article 35.

Exclusion Criteria:

1. Any maternal or fetal contraindication to vaginal delivery
2. Known uterine anomaly
3. Multifetal gestation
4. Estimated fetal weight of 4500 gm or greater
5. Ruptured membranes

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 204 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Bliss, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Six Hour | Twelve Hour
Started | 103 | 101
Completed | 101 | 99
Not Completed | 2 | 2
Not completed — Screen Failure | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Six Hour | Twelve Hour | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.8 (5.96) | 24.33 (5.92) | 24.6 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 99 | 200
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 49 | 42 | 91
  White | 16 | 18 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 35 | 35 | 70
Maternal Weight [Mean (Standard Deviation); unit: kg] | 89.0 (20.6) | 85.9 (19.0) | 87.5 (19.8)
Maternal BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.1 (7.5) | 32.7 (6.6) | 33.4 (7.1)
Gestational Age [Mean (Standard Deviation); unit: wks] | 39.4 (1.4) | 39.5 (1.4) | 39.5 (1.4)
Gravidity [Mean (Standard Deviation); unit: events] | 1.4 (0.9) | 1.4 (0.7) | 1.4 (0.8)
Parity [Mean (Standard Deviation); unit: Events] | 0.1 (0.3) | 0.1 (0.4) | 0.1 (0.4)
Bishop score on admission [Mean (Standard Deviation); unit: Score] — The Bishop score is used to rate the readiness of the cervix for labor. Score ranges from 0 to 13. A Bishop score of less than 6 means that the cervix may not be ready for labor.
  Score | 3.1 (1.5) | 3.2 (1.5) | 3.2 (1.5)
Indication for Induction [Count of Participants; unit: Participants]
  Postdates | 23 | 23 | 46
  Oligohydramnios | 8 | 11 | 19
  Maternal Health Condition | 62 | 53 | 115
  Fetal Health Condition | 16 | 22 | 38
  Other | 3 | 3 | 6
concomitant medications during induction [Count of Participants; unit: Participants]
  Magnesium Sulfate | 20 | 12 | 32
  Pitocin w Foley Bulb | 14 | 14 | 28
  Pitocin after Foley Bulb | 97 | 94 | 191
  Misoprostol prior to Foley Bulb | 35 | 27 | 62
  Misoprostol w Foley Bulb | 1 | 2 | 3
  Epidural | 97 | 97 | 194

OUTCOME MEASURES:

1. Primary Outcome: Time From Foley Bulb Placement to Time of Delivery.
Description: Time in hours to delivery following use of foley catheter
Time Frame: Change in time to delivery following bulb insertion for 6 hours up to 72 hours
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
hr | 24.2 (10.2) | 24.57 (10.1)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.8, t-test, 2 sided

2. Primary Outcome: Time to Delivery of Trial of Labor After Cesarean Section
Time Frame: Time (hours) to delivery
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 13 | 11
hours | 20.62 (8.8) | 27.18 (11.9)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.133, t-test, 2 sided

3. Primary Outcome: 1 Minute Apgar Score of Trial of Labor After Cesarean Section
Description: The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
Time Frame: 1 minute Apgar score following birth
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 13 | 11
score on a scale | 7.6 (2.4) | 7.3 (2.3)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.58, t-test, 2 sided

4. Secondary Outcome: Time From Foley Bulb Placement to Extrusion
Description: Time in hours from foley bulb placement to extrusion
Time Frame: Hour 6, Hour 12
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
hrs | 5.75 (0.9) | 9.25 (3.5)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mode of Delivery--Number of Participants Having Cesarean Delivery
Time Frame: Hour Six, Hour 12
Measure: Count of Participants; unit: Participants
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
Participants | 34 | 35
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.8, Chi-squared

6. Secondary Outcome: Bacterial Infection (Chorioamnionitis)
Time Frame: Hour Six, Hour 12
Measure: Count of Participants; unit: Participants
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
Participants | 16 | 16
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.95, Chi-squared

7. Secondary Outcome: Endometritis
Time Frame: Hour 6, Hour 12
Measure: Count of Participants; unit: Participants
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
Participants | 4 | 4
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.98, Chi-squared

8. Secondary Outcome: 1 Minute Apgar Score
Description: as for outcome 3
Time Frame: 1 minute Apgar score following birth
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
Score | 8 (1.8) | 7.9 (1.9)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.95, t-test, 2 sided

9. Secondary Outcome: 5 Minute Apgar Score
Description: as for outcome 3
Time Frame: 5 minute Apgar score following birth
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 101 | 99
Score | 8.8 (0.7) | 8.8 (1.0)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.1, t-test, 2 sided

10. Secondary Outcome: Time to Foley Bulb Extrusion of Trial of Labor After Cesarean Section
Time Frame: Time to foley bulb extrusion
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 13 | 11
hours | 5.6 (1.0) | 10.6 (3.1)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.0003, t-test, 2 sided

11. Secondary Outcome: 5 Minute Apgar Score of Trial of Labor After Cesarean Section
Description: as for outcome 3
Time Frame: 5 Minute Apgar Score following birth
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Six Hour | Twelve Hour
Number analyzed (Participants) | 13 | 11
score on a scale | 8.7 (0.6) | 8.4 (2.1)
Statistical Analysis 1: Comparison: Six Hour vs Twelve Hour; Test type: Superiority; p = 0.48, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Six Hour | Twelve Hour
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99
Other Adverse Events (participants affected / at risk) | 0/101 | 1/99
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Six Hour (N=101) | Twelve Hour (N=99)
incorrect foley placement (Pregnancy, puerperium and perinatal conditions) | 0 | 1 — foley bulb was not placed in the cervix

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes